CLINICAL TRIAL: NCT07205367
Title: Validation Study: Extended Wear Performance of the Zio Monitor - SHASTA II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: iRhythm Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: iRT-003-2024
Record Dates: First submitted 2025-09-09; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: This is a design validation study to evaluate the wear performance of the Zio monitor/Zio MCT device form factor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Open Label (Other): This is an open-label study. All participants will have the study device applied to their chest. Two-thirds of the participants will have the study device applied by a Study Staff member (i.e., Healthcare Provider (HCP)). One-third of the participants will self-apply the study device to their chest (i.e., simulated at-home patch application). Application of all study devices will be performed at the site.
  Interventions: Device: Zio Monitor

INTERVENTIONS:
Device: Zio Monitor — The Zio monitor is a long-term continuous ambulatory patch ECG monitor which adheres to the patient's left pectoral region.

SUMMARY:
This trial assesses the wear performance of the Zio monitor, a long-term continuous ambulatory patch ECG monitor, in a representative population by evaluating (1) the wear duration (up to 30 days) of the device, (2) the percentage of analyzable electrocardiographic time and (3) safety by reviewing all adverse events.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm study to validate the design of the Zio monitor/Zio MCT device form factor in extended (21-day) wear when utilizing an updated skin prep process.

The trial is conducted in 2 phases. Phase I includes the standard skin preparation process of 40 strokes with an exfoliator in 4 different directions. Phase II incorporates a modified skin preparation process: only 20 strokes with an exfoliator in 2 directions are used. There are 75 participants in each phase.

Performance objectives include the following: (1) Mean wear duration of 21 days and (2) percent analyzable time of 80%.

Safety measures include the proportion of participants that experience clinically significant skin irritation through 30 days of wear, as well as the reporting of all adverse events.

Additional device measures include the following: (1) % signal artifact (defined as the proportion of ECG signal that is artifact over the wear duration, reported for each study device); (2) % device functionality (defined as the proportion of Zio monitors recording a continuous ECG signal through 21 days, and through 30 days) and (3) observational assessment of participant skin types (assessed by dryness levels, hyperhydrosis status, Fitzpatrick Skin Type and chest hair density).

All analyses will be performed on the population of enrolled participants on whom the Zio monitor application was attempted. The age, sex at birth, and application type (i.e., healthcare provider (HCP) designee vs. self-application) of participants will be monitored throughout the enrollment period to ensure representation across key user groups. Performance within subgroups including (but not limited to) sex at birth, age, and application type will be assessed.

Up to 150 participants will be enrolled at 2 US iRhythm locations (San Francisco, CA and Deerfield, IL).

There are 3 on-location visits at Baseline (Visit 1/time of patch application), Day 21 (Visit 4) and Day 30 (Visit 5/following 30 days of patch application). There are 2 telephone/video calls at Day 7 (Visit 2) and Day 14 (Visit 3).

Participants who meet all inclusion criteria and no exclusion criteria will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 years or older at time of informed consent.
2. Participant is willing and able to provide informed consent and be able to complete all visits for the study.

Exclusion Criteria:

1. Participant has a known allergy to adhesives.
2. Participant has a current skin infection or injury at location for study device placement.
3. Participant is a member of a vulnerable population.
4. Participant is a current or prior employee of iRhythm.
5. Participant is unable or unwilling to participate or comply with study protocol.
6. The local Investigator deems the participant has a condition that could limit the participant's ability or willingness to participate in the study, or ability to comply with study required procedures and/or follow-up visits.
7. Participant has experienced symptomatic episodes where instance variations in cardiac performance could result in immediate danger to the participant.
8. Participant has an external cardiac defibrillator or may be exposed to high frequency surgical equipment near strong magnetic fields or devices such as MRI during the wear period.
9. Participant has a neuro-stimulator, as it may disrupt the quality of ECG data.
10. Participant does not have the competency to wear the device for the prescribed monitoring period.
11. Participant does not have the ability to consent for themselves (i.e., no LARs).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Mean Wear Duration | 21 - 30 days after baseline
  This outcome measure is met if the mean wear duration is greater than 21 days
Percent Analyzable Time | Up to 30 days (Day 30)
  This outcome measure is met if the percent analyzable time is greater than 80% in 90% of subjects.
Safety: Skin Irritation | Up to 30 days (Day 30)
  This includes the proportion of participants that experience clinically significant skin irritation through 30 days of wear. This will be assessed through the capture and reporting of all adverse events

SECONDARY OUTCOMES:
Additional Device Measure 1: Percent Signal Artifact | Up to 30 days (Day 30)
  Percent signal artifact is defined as the proportion of ECG signal that is artifact over the wear duration, reported for each study device.
Additional Device Measure 2: Percent Device Functionality | At 21 days (Day 21) and 30 days (Day 30)
  Percent device functionality is defined as the proportion of Zio monitors recording a continuous ECG signal through 21 days, and through 30 days.
Observational Assessment: Skin Dryness Level | Baseline (Day 1)
  This includes an assessment of the following skin types: dry, oily and normal.
Observational Assessment: Hyperhydrosis Status | Baseline (Day 1)
  This includes an assessment of the following hyperhydrosis status: primary, secondary or none.
Observational Assessment: Fitzpatrick Skin Type | Baseline (Day 1)
  This includes a 6-point scale to assess the following skin types: (1) pale skin; always burns, never tans; (2) fair skin; usually burns, tans minimally; (3) darker white skin; sometimes mild burn, tans uniformly; (4) light brown skin; burns minimally, always tans well; (5) brown skin; very rarely burns; tans very easily; (6) dark brown or black skin; never burns.
Observational Assessment: Chest Hair Density | Baseline (Day 1), 21 days (Day 21) and 30 days (Day 30)
  This includes an assessment of the following chest hair density types: smooth/no hair; some hair; moderately hairy; or very hairy in the target patch placement area.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - iRhythm Technologies - San Francisco, CA, San Francisco, California
  - iRhythm Technologies - Deerfield, IL, Deerfield, Illinois

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.

DOCUMENTS (1):
  • Study Protocol (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT07205367/Prot_000.pdf